CLINICAL TRIAL: NCT00937859
Title: A Phase III Randomized, Double Blind, Placebo Control, Multicenter Study to Investigate the Efficacy and Safety of SER120 Nasal Spray Formulation in Patients With Nocturia
Brief Title: Treatment of Patients With Nocturia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Serenity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPC-SER120-DB1-200901
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Results first posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2014-04

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SER120 (Experimental): SER120
  Interventions: Drug: SER120
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SER120 — SER120
  Arms: SER120
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate a treatment of nocturia. The hypothesis is that SER120 will decrease the number of nocturic episodes compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and female 50 years or older
* Nocturia of 6 or more months duration averaging 2 episodes or more per night

Exclusion Criteria:

* CHF
* Diabetes
* Diabetes Insipidus
* Renal Insufficiency
* Hepatic Insufficiency
* Incontinence
* Illness requiring steroids
* Current or past urologic malignancy
* Nephrotic Syndrome
* Unexplained pelvic masses
* Urinary bladder neurological dysfunction
* Urinary bladder surgery or radiotherapy
* Sleep Apnea
* Pregnant or breast feeding

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Piedmont Medical Research Assoc., Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SER120: All participants received SER120 500 ng once daily for at least 1 week and, if needed, participants were allowed to up-titrate to SER120 750 ng once daily for the remainder of the study.
- Placebo: All participants received placebo once daily for at least 1 week and were allowed to undergo a mock up-titration once daily for the remainder of the study.
Period: Overall Study
Arm/Group | SER120 | Placebo
Started | 148 | 153
Completed | 129 | 134
Not Completed | 19 | 19

BASELINE CHARACTERISTICS:
Population: Intent-to-treat
Groups:
- Placebo: All participants received placebo once daily for at least 1 week and were allowed to undergo a mock up-titration with placebo once daily for the remainder of the study.
- Total: Total of all reporting groups
Arm/Group | SER120 | Placebo | Total
Number analyzed (Participants) | 145 | 149 | 294
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (9.4) | 63.7 (9.6) | 63.7 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 62 | 128
  Male | 79 | 87 | 166
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 8 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 23 | 42
  White | 121 | 115 | 236
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 145 | 149 | 294

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Number of Nocturic Episodes/Night
Description: Change was calculated as the mean number of nocturic episodes per night during the last week of treatment minus the mean number of nocturic episodes at baseline
Time Frame: 7 weeks
Population: Intent-to-treat
Measure: Least Squares Mean (Standard Deviation); unit: nocturic episodes per night
Arm/Group | SER120 | Placebo
Number analyzed (Participants) | 145 | 149
nocturic episodes per night | -1.3 (0.9) | -1.2 (1.0)

2. Primary Outcome: Percent of Participants With at Least 50% Decrease in Mean Nocturic Episodes Per Night
Description: Percent of participants achieving at least 50% reduction in nocturic episodes during the last week of treatment compared to baseline
Time Frame: 7 weeks
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | SER120 | Placebo
Number analyzed (Participants) | 145 | 149
Participants | 58 | 58

ADVERSE EVENTS:
Arm/Group | SER120 | Placebo
Serious Adverse Events (participants affected / at risk) | 2/148 | 1/153
Other Adverse Events (participants affected / at risk) | 105/148 | 108/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SER120 (N=148) | Placebo (N=153)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SER120 (N=148) | Placebo (N=153)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 7 (7)
Nasopharyngitis (Infections and infestations) | 7 (7) | 4 (4)
Headache (Nervous system disorders) | 6 (6) | 16 (16)
Dizziness (Nervous system disorders) | 2 (2) | 7 (7)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 44 (44) | 58 (58)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 22 (22)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 22 (22)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (8)
throat irritation (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Post nasal drip (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes